CLINICAL TRIAL: NCT04104685
Title: A Prospective, Multicenter, Randomized, Double-Blind, Vehicle-Controlled Phase 2 Study to Evaluate the Safety and Efficacy of a Combination of 3% Minocycline and 0.3% Adapalene Topical Foam Formulation for the Treatment of Moderate-to-Severe Acne (Study FX2016 40)
Brief Title: A Study to Compare FCD105 Foam to Minocycline 3% Foam, Adapalene 0.3% Foam and Vehicle Foam.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FX2016-40
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- FCD105 Foam (Experimental): FCD105 Foam
  Interventions: Combination Product: FCD105
- 3% Minocycline Foam (Active Comparator): 3% Minocycline Foam
  Interventions: Drug: 3% Minocycline Foam
- 0.3% Adapalene Foam (Active Comparator): 0.3% Adapalene Foam
  Interventions: Drug: 0.3% Adapalene Foam
- Vehicle Foam (Placebo Comparator): Vehicle Foam
  Interventions: Other: Vehicle Foam

INTERVENTIONS:
Combination Product: FCD105 — Experimental combination
  Arms: FCD105 Foam
Drug: 3% Minocycline Foam — Active Comparator
  Arms: 3% Minocycline Foam
Drug: 0.3% Adapalene Foam — Active Comparator
  Arms: 0.3% Adapalene Foam
Other: Vehicle Foam — Placebo
  Arms: Vehicle Foam

SUMMARY:
A study comparing FCD105 to 3% minocycline foam, 0.3% adapalene foam and vehicle foam in patients ≥ 12 years old for the treatment of moderate-to-severe acne.

ELIGIBILITY:
Inclusion Criteria:

1. Has facial acne vulgaris with all of the following:

   1. 20 to 50 inflammatory lesions (papules and/or pustules) on the face.
   2. 25 to 100 non-inflammatory lesions (open and closed comedones) on the face.
   3. IGA score of moderate (3) to severe (4).
2. No more than two active nodules on the face.
3. Willing to use only the supplied non-medicated cleanser and to refrain from use of any other acne medication, medicated cleanser, excessive sun exposure, and tanning booths for the duration of the study

Exclusion Criteria:

1. Female who is pregnant or lactating, or is planning a pregnancy during the study.
2. Acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne), or any dermatological condition of the face that could interfere with the clinical evaluations.
3. Facial hair (eg, beard, mustache, etc.) that could interfere with the clinical evaluations.
4. Sunburn on the face.
5. Severe systemic disease as assessed by the Investigator that might interfere with the conduct of the study or the interpretation of the results.
6. Subjects who have a documented history of any of the following:

   1. Allergy to tetracycline-class antibiotics or to any ingredient in the study drug.
   2. Pseudomembranous colitis or antibiotic-associated colitis.
   3. Hepatitis or clinically significant liver damage or clinically significant renal impairment.
   4. Known or suspected premalignant or malignant disease (excluding successfully treated skin cancers).
7. Subjects who have used the following medications:

   Within 1 week prior to randomization:
   * Medicated facial cleansers on the face.
   * Topical acne treatments on the face (other than those listed below).

   Within 4 weeks prior to randomization:
   * Topical retinoids on the face.
   * Topical anti-inflammatories and/or corticosteroids on the face.
   * Topical corticosteroids on body areas other than the face for more than 15 consecutive days and on more than 10% of the body surface area. In body folds, such as axillary and inguinal regions, only mild topical steroids are allowed for short term use (≤15 consecutive days).
   * Systemic antibiotics.
   * Systemic acne treatments.

   Within 12 weeks prior to randomization:
   * Systemic retinoids.
   * Systemic corticosteroids (Note: Intranasal and inhaled corticosteroids may be used throughout the study if the subject is on a stable dose).
8. Use of sauna during the 2 weeks prior to randomization.
9. Epilation of the face within 2 weeks prior to randomization.
10. Folliculitis on the face.
11. Documented history of depression that is not, in the opinion of the Investigator, currently adequately controlled with medication

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Absolute change from Baseline in inflammatory lesion counts at week 12 | 12 weeks
  Statistical superiority of FCD105 vs. vehicle in the absolute change from Baseline in inflammatory lesion counts at Visit 4 (Week12/End of Treatment)
Absolute change from Baseline in non-inflammatory lesion counts at week 12 | 12 weeks
  Statistical superiority of FCD105 vs. vehicle in the absolute change from Baseline in non-inflammatory lesion counts at Visit 4 (Week12/End of Treatment)
Investigator's Global Assessment (IGA) Treatment Success at Week 12 | 12 weeks
  Statistical superiority of FCD105 vs. vehicle in in IGA Treatment Success at Visit 4 (Week 12/End of Treatment), where success is defined as an IGA score of 0 or 1, and at least a 2-grade improvement (decrease) from Baseline.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Foamix Institution #134, Bryant, Arkansas
  - Foamix Institution #121, Rogers, Arkansas
  - Foamix Institution #106, Encino, California
  - Foamix Institution #103, Fremont, California
  - Foamix Institution #122, Huntington Beach, California
  - Foamix Institution #109, Manhattan Beach, California
  - Foamix Institution #132, San Diego, California
  - Foamix Institution #107, Hialeah, Florida
  - Foamix Institution #127, Lake City, Florida
  - Foamix Institution #101, Miami, Florida
  - Foamix Institution #135, Miami Beach, Florida
  - Foamix Institution #118, Sanford, Florida
  - Foamix Institution #120, Sunrise, Florida
  - Foamix Institution #128, Tampa, Florida
  - Foamix Institution #130, New Albany, Indiana
  - Foamix Institution #116, Plainfield, Indiana
  - Foamix Institution #123, Louisville, Kentucky
  - Foamix Institution #126, Baton Rouge, Louisiana
  - Foamix Institution #124, New Orleans, Louisiana
  - Foamix Institution #136, Watertown, Massachusetts
  - Foamix Institution #114, Clinton Township, Michigan
  - Foamix Institution #111, Fridley, Minnesota
  - Foamix Institution #102, Las Vegas, Nevada
  - Foamix Institution #115, New York, New York
  - Foamix Institution #108, Stony Brook, New York
  - Foamix Institution #104, High Point, North Carolina
  - Foamix Institution #133, Gresham, Oregon
  - Foamix Institution #125, Johnston, Rhode Island
  - Foamix Institution #119, Mt. Pleasant, South Carolina
  - Foamix Institution #110, Arlington, Texas
  - Foamix Institution #117, College Station, Texas
  - Foamix Institution #112, Pflugerville, Texas
  - Foamix Institution #105, San Antonio, Texas
  - Foamix Institution #131, Layton, Utah
  - Foamix Institution #113, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No